CLINICAL TRIAL: NCT05609266
Title: Validation of Non-invasive Risk Models for Prediction of Incident Type 2 Diabetes in a Swedish Population
Brief Title: Validation of Existing Diabetes Risk Models in a Swedish Population
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-VIPRisk_Valexist
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Type2diabetes
Keywords: Non-invasive prediction model; Incident diabetes; Validation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to validate existing non-invasive diabetes clinical prediction models in a Swedish population. The main question it aims to answer is: how well 11 existing models will perform in predicting incident type 2 diabetes in participants from the Västerbotten Intervention programme (VIP). Participants in VIP are residents of Västerbotten that are invited for a comprehensive health screening at 30- (until 1995), 40-, 50-, and 60-years of age.

DETAILED DESCRIPTION:
Several type 2 diabetes risk prediction models have been developed but how it will perform in a Swedish population is not known. No diabetes risk prediction model is routinely used in Sweden. The aim of this study is therefore, to validate 11 non-invasive models and to evaluate the performance to predict incident type 2 diabetes in a Swedish population. A population-based cohort from the Västerbotten Intervention programme (VIP) from 1990 to 2020 will be the validation sample. Incident type 2 diabetes within 10-years of follow-up, will be determined by oral glucose tolerance test or through self-reports. A self-administered questionnaire is completed, and anthropometric, clinical, and biochemical measures are obtained at each of the health screening visits. In the statistical analysis the overall performance of the models will be compared using the Brier score. In addition. discrimination and calibration of all the models will be evaluated. Recalibration of models will be done.

ELIGIBILITY:
Inclusion Criteria:

• At least one visit within the Västerbotten Intervention program

Exclusion Criteria:

• Prevalent diabetes at first visit defined by a fasting capillary plasma glucose >7mmol/L, a 2-hour capillary plasma glucose of ≥12.2 mmol/L or self-reported history of diabetes

Ages: 28 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Inhabitants from the Västerbotten region in Sweden that have been invited to participate in the Västerbotten Intervention Program for a comprehensive health screening at 30 (stopped in 1995) 40, 50 and 60 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 115642 (Actual)
Dates: Start 1990-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Incident type 2 diabetes | 10-years
  Determined by a fasting capillary plasma glucose of ≥7 mmol/L or a 2-hour capillary plasma glucose of ≥12.2 mmol/L, or self-reported

CONTACTS AND LOCATIONS:
Overall Officials: Olov Rolandsson, MD, Principal Investigator — Umeå University

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available due to the protection of privacy and data sharing constraints. Applications to access the data may be submitted to the Biobank Research Unit at Umeå University.

REFERENCES:
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Background] Cho NH, Shaw JE, Karuranga S, Huang Y, da Rocha Fernandes JD, Ohlrogge AW, Malanda B. IDF Diabetes Atlas: Global estimates of diabetes prevalence for 2017 and projections for 2045. Diabetes Res Clin Pract. 2018 Apr;138:271-281. doi: 10.1016/j.diabres.2018.02.023. Epub 2018 Feb 26. PMID 29496507
- [Background] Li G, Zhang P, Wang J, Gregg EW, Yang W, Gong Q, Li H, Li H, Jiang Y, An Y, Shuai Y, Zhang B, Zhang J, Thompson TJ, Gerzoff RB, Roglic G, Hu Y, Bennett PH. The long-term effect of lifestyle interventions to prevent diabetes in the China Da Qing Diabetes Prevention Study: a 20-year follow-up study. Lancet. 2008 May 24;371(9626):1783-9. doi: 10.1016/S0140-6736(08)60766-7. PMID 18502303
- [Background] Gillies CL, Abrams KR, Lambert PC, Cooper NJ, Sutton AJ, Hsu RT, Khunti K. Pharmacological and lifestyle interventions to prevent or delay type 2 diabetes in people with impaired glucose tolerance: systematic review and meta-analysis. BMJ. 2007 Feb 10;334(7588):299. doi: 10.1136/bmj.39063.689375.55. Epub 2007 Jan 19. PMID 17237299
- [Background] Simmons RK, Griffin SJ, Lauritzen T, Sandbaek A. Effect of screening for type 2 diabetes on risk of cardiovascular disease and mortality: a controlled trial among 139,075 individuals diagnosed with diabetes in Denmark between 2001 and 2009. Diabetologia. 2017 Nov;60(11):2192-2199. doi: 10.1007/s00125-017-4299-y. Epub 2017 Aug 23. PMID 28831539
- [Background] Herman WH, Ye W, Griffin SJ, Simmons RK, Davies MJ, Khunti K, Rutten GE, Sandbaek A, Lauritzen T, Borch-Johnsen K, Brown MB, Wareham NJ. Early Detection and Treatment of Type 2 Diabetes Reduce Cardiovascular Morbidity and Mortality: A Simulation of the Results of the Anglo-Danish-Dutch Study of Intensive Treatment in People With Screen-Detected Diabetes in Primary Care (ADDITION-Europe). Diabetes Care. 2015 Aug;38(8):1449-55. doi: 10.2337/dc14-2459. Epub 2015 May 18. PMID 25986661
- [Background] Sortso C, Komkova A, Sandbaek A, Griffin SJ, Emneus M, Lauritzen T, Simmons RK. Effect of screening for type 2 diabetes on healthcare costs: a register-based study among 139,075 individuals diagnosed with diabetes in Denmark between 2001 and 2009. Diabetologia. 2018 Jun;61(6):1306-1314. doi: 10.1007/s00125-018-4594-2. Epub 2018 Mar 16. PMID 29549417
- [Background] Kengne AP, Beulens JW, Peelen LM, Moons KG, van der Schouw YT, Schulze MB, Spijkerman AM, Griffin SJ, Grobbee DE, Palla L, Tormo MJ, Arriola L, Barengo NC, Barricarte A, Boeing H, Bonet C, Clavel-Chapelon F, Dartois L, Fagherazzi G, Franks PW, Huerta JM, Kaaks R, Key TJ, Khaw KT, Li K, Muhlenbruch K, Nilsson PM, Overvad K, Overvad TF, Palli D, Panico S, Quiros JR, Rolandsson O, Roswall N, Sacerdote C, Sanchez MJ, Slimani N, Tagliabue G, Tjonneland A, Tumino R, van der A DL, Forouhi NG, Sharp SJ, Langenberg C, Riboli E, Wareham NJ. Non-invasive risk scores for prediction of type 2 diabetes (EPIC-InterAct): a validation of existing models. Lancet Diabetes Endocrinol. 2014 Jan;2(1):19-29. doi: 10.1016/S2213-8587(13)70103-7. Epub 2013 Oct 8. PMID 24622666
- [Background] Balkau B, Lange C, Fezeu L, Tichet J, de Lauzon-Guillain B, Czernichow S, Fumeron F, Froguel P, Vaxillaire M, Cauchi S, Ducimetiere P, Eschwege E. Predicting diabetes: clinical, biological, and genetic approaches: data from the Epidemiological Study on the Insulin Resistance Syndrome (DESIR). Diabetes Care. 2008 Oct;31(10):2056-61. doi: 10.2337/dc08-0368. Epub 2008 Aug 8. PMID 18689695
- [Background] Chen L, Magliano DJ, Balkau B, Colagiuri S, Zimmet PZ, Tonkin AM, Mitchell P, Phillips PJ, Shaw JE. AUSDRISK: an Australian Type 2 Diabetes Risk Assessment Tool based on demographic, lifestyle and simple anthropometric measures. Med J Aust. 2010 Feb 15;192(4):197-202. doi: 10.5694/j.1326-5377.2010.tb03507.x. PMID 20170456
- [Background] Griffin SJ, Little PS, Hales CN, Kinmonth AL, Wareham NJ. Diabetes risk score: towards earlier detection of type 2 diabetes in general practice. Diabetes Metab Res Rev. 2000 May-Jun;16(3):164-71. doi: 10.1002/1520-7560(200005/06)16:33.0.co;2-r. PMID 10867715
- [Background] Lindstrom J, Tuomilehto J. The diabetes risk score: a practical tool to predict type 2 diabetes risk. Diabetes Care. 2003 Mar;26(3):725-31. doi: 10.2337/diacare.26.3.725. PMID 12610029
- [Background] Hippisley-Cox J, Coupland C, Robson J, Sheikh A, Brindle P. Predicting risk of type 2 diabetes in England and Wales: prospective derivation and validation of QDScore. BMJ. 2009 Mar 17;338:b880. doi: 10.1136/bmj.b880. PMID 19297312
- [Background] Rahman M, Simmons RK, Harding AH, Wareham NJ, Griffin SJ. A simple risk score identifies individuals at high risk of developing Type 2 diabetes: a prospective cohort study. Fam Pract. 2008 Jun;25(3):191-6. doi: 10.1093/fampra/cmn024. Epub 2008 May 30. PMID 18515811
- [Background] Rosella LC, Manuel DG, Burchill C, Stukel TA; PHIAT-DM team. A population-based risk algorithm for the development of diabetes: development and validation of the Diabetes Population Risk Tool (DPoRT). J Epidemiol Community Health. 2011 Jul;65(7):613-20. doi: 10.1136/jech.2009.102244. Epub 2010 Jun 1. PMID 20515896
- [Background] Schmidt MI, Duncan BB, Bang H, Pankow JS, Ballantyne CM, Golden SH, Folsom AR, Chambless LE; Atherosclerosis Risk in Communities Investigators. Identifying individuals at high risk for diabetes: The Atherosclerosis Risk in Communities study. Diabetes Care. 2005 Aug;28(8):2013-8. doi: 10.2337/diacare.28.8.2013. PMID 16043747
- [Background] Schulze MB, Hoffmann K, Boeing H, Linseisen J, Rohrmann S, Mohlig M, Pfeiffer AF, Spranger J, Thamer C, Haring HU, Fritsche A, Joost HG. An accurate risk score based on anthropometric, dietary, and lifestyle factors to predict the development of type 2 diabetes. Diabetes Care. 2007 Mar;30(3):510-5. doi: 10.2337/dc06-2089. PMID 17327313
- [Background] Abbasi A, Peelen LM, Corpeleijn E, van der Schouw YT, Stolk RP, Spijkerman AM, van der A DL, Moons KG, Navis G, Bakker SJ, Beulens JW. Prediction models for risk of developing type 2 diabetes: systematic literature search and independent external validation study. BMJ. 2012 Sep 18;345:e5900. doi: 10.1136/bmj.e5900. PMID 22990994
- [Background] Wilson PW, Meigs JB, Sullivan L, Fox CS, Nathan DM, D'Agostino RB Sr. Prediction of incident diabetes mellitus in middle-aged adults: the Framingham Offspring Study. Arch Intern Med. 2007 May 28;167(10):1068-74. doi: 10.1001/archinte.167.10.1068. PMID 17533210
- [Background] Kahn HS, Cheng YJ, Thompson TJ, Imperatore G, Gregg EW. Two risk-scoring systems for predicting incident diabetes mellitus in U.S. adults age 45 to 64 years. Ann Intern Med. 2009 Jun 2;150(11):741-51. doi: 10.7326/0003-4819-150-11-200906020-00002. PMID 19487709
- [Background] Collins GS, Mallett S, Omar O, Yu LM. Developing risk prediction models for type 2 diabetes: a systematic review of methodology and reporting. BMC Med. 2011 Sep 8;9:103. doi: 10.1186/1741-7015-9-103. PMID 21902820
- [Background] Collins GS, Reitsma JB, Altman DG, Moons KG. Transparent reporting of a multivariable prediction model for individual prognosis or diagnosis (TRIPOD): the TRIPOD Statement. BMC Med. 2015 Jan 6;13:1. doi: 10.1186/s12916-014-0241-z. PMID 25563062
- [Background] Moons KG, Altman DG, Reitsma JB, Ioannidis JP, Macaskill P, Steyerberg EW, Vickers AJ, Ransohoff DF, Collins GS. Transparent Reporting of a multivariable prediction model for Individual Prognosis or Diagnosis (TRIPOD): explanation and elaboration. Ann Intern Med. 2015 Jan 6;162(1):W1-73. doi: 10.7326/M14-0698. PMID 25560730
- [Background] Norberg M, Wall S, Boman K, Weinehall L. The Vasterbotten Intervention Programme: background, design and implications. Glob Health Action. 2010 Mar 22;3. doi: 10.3402/gha.v3i0.4643. PMID 20339479
- [Background] Norberg M, Blomstedt Y, Lonnberg G, Nystrom L, Stenlund H, Wall S, Weinehall L. Community participation and sustainability--evidence over 25 years in the Vasterbotten Intervention Programme. Glob Health Action. 2012 Dec 17;5:1-9. doi: 10.3402/gha.v5i0.19166. PMID 23528041
- [Background] Feldman AL, Griffin SJ, Fharm E, Norberg M, Wennberg P, Weinehall L, Rolandsson O. Screening for type 2 diabetes: do screen-detected cases fare better? Diabetologia. 2017 Nov;60(11):2200-2209. doi: 10.1007/s00125-017-4402-4. Epub 2017 Aug 23. PMID 28831538
- [Background] Chen Y, Copeland WK, Vedanthan R, Grant E, Lee JE, Gu D, Gupta PC, Ramadas K, Inoue M, Tsugane S, Tamakoshi A, Gao YT, Yuan JM, Shu XO, Ozasa K, Tsuji I, Kakizaki M, Tanaka H, Nishino Y, Chen CJ, Wang R, Yoo KY, Ahn YO, Ahsan H, Pan WH, Chen CS, Pednekar MS, Sauvaget C, Sasazuki S, Yang G, Koh WP, Xiang YB, Ohishi W, Watanabe T, Sugawara Y, Matsuo K, You SL, Park SK, Kim DH, Parvez F, Chuang SY, Ge W, Rolland B, McLerran D, Sinha R, Thornquist M, Kang D, Feng Z, Boffetta P, Zheng W, He J, Potter JD. Association between body mass index and cardiovascular disease mortality in east Asians and south Asians: pooled analysis of prospective data from the Asia Cohort Consortium. BMJ. 2013 Oct 1;347:f5446. doi: 10.1136/bmj.f5446. PMID 24473060
- [Background] Lee KJ, Carlin JB. Multiple imputation for missing data: fully conditional specification versus multivariate normal imputation. Am J Epidemiol. 2010 Mar 1;171(5):624-32. doi: 10.1093/aje/kwp425. Epub 2010 Jan 27. PMID 20106935
- [Background] White IR, Royston P, Wood AM. Multiple imputation using chained equations: Issues and guidance for practice. Stat Med. 2011 Feb 20;30(4):377-99. doi: 10.1002/sim.4067. Epub 2010 Nov 30. PMID 21225900
- [Background] Steyerberg EW, Vickers AJ, Cook NR, Gerds T, Gonen M, Obuchowski N, Pencina MJ, Kattan MW. Assessing the performance of prediction models: a framework for traditional and novel measures. Epidemiology. 2010 Jan;21(1):128-38. doi: 10.1097/EDE.0b013e3181c30fb2. PMID 20010215
- See also: WHO Definition, diagnosis and classification of diabetes mellitus and its complications — https://apps.who.int/iris/handle/10665/66040